CLINICAL TRIAL: NCT01824004
Title: A Phase II Study of Adjuvant S-1/Cisplatin Chemotherapy Followed by S-1-based Chemoradiotherapy in Advanced Gastric Cancer
Brief Title: Postoperative Chemoradiotherapy With S-1 in Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chonnam National University Hospital (Other)
Responsible Party: Principal Investigator, Sang-Hee Cho, Professor, Chonnam National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNUHH-MO-03; CNUHH (Other Grant/Funding Number: Jeil Pham)
Record Dates: First submitted 2013-03-28; First posted 2013-04-04 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Gastric Cancer
Keywords: Gastric cancer; Adjuvant; Chemoradiotherapy; S-1; Cisplatin
MeSH Terms: conditions — Stomach Neoplasms | interventions — S 1 (combination); titanium silicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- S-1,chemoradiotherapy, adjuvant treatment (Experimental): Pts with radically D2 resected adenocarcinoma of the stomach or GEJ in AJCC stage Ib-IV (M0) were eligible for this study. Pts were treated with S-1 (40-60 mg depending on BSA) b.i.d. for 3 wks, and cisplatin (60 mg/m²) iv on day 1, followed by a 2-wk rest period, within a 5-wk cycle. Subsequently, radiotherapy (RT) started which consisted of 25 fractions of 1.8 Gy to a total dose of 45 Gy in 5 wks (5 fractions/wk). On RT days, S-1 (40-60 mg depending on BSA ) b.i.d., 5 days/wk was given. One month after the completion of RT, two 5-wk cycles of S-1/ciplatin chemotherapy were given.
  Interventions: Drug: S-1

INTERVENTIONS:
Drug: S-1
  Other Names: TS-1

SUMMARY:
This study was conducted to evaluate the clinical outcomes and toxicities of adjuvant treatment including S-1/cisplatin chemotherapy followed by S-1 based CRT.

DETAILED DESCRIPTION:
Surgery is the only possible curative treatment of gastric cancer. However, the high recurrence rate makes gastric cancer a disease difficult to cure by surgery alone. Despite the benefit of CRT on local recurrence, the distant recurrence is the leading pattern of failure. We hypothesized that gastric cancer outcome could be improved using a more effective chemotherapy regimen. This study was conducted to evaluate the clinical outcomes and toxicity of adjuvant treatment including S-1/cisplatin chemotherapy followed by S-1 based CRT.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Histologically proven gastric adenocarcinoma which is complete resected
* ECOG performance status of 1 or lower
* Adequate bone marrow function

  * absolute neutrophil count [ANC] ≥1,500µL, and platelets ≥100,000/µL
* Adequate kidney function (serum creatinine < 1.5 mg/dL)
* Adequate liver function (serum total bilirubin < 2 times the upper normal limit (UNL) serum transaminases levels <2 times UNL
* No prior chemotherapy

Exclusion Criteria:

* Other tumor type than adenocarcinoma
* Evidence of distant metastasis
* Past or concurrent history of neoplasm except for curatively treated non-melanoma skin cancer or in situ carcinoma of the cervix uteri
* Uncontrolled infection
* Unstable cardiac disease despite treatment, myocardial infarction within months prior to study entry
* History of significant neurologic or psychiatric disorders including dementia or seizures
* Other serious underlying medical conditions which could impair the ability of the patient to participate in the study
* Symptoms of gastrointestinal obstruction
* concomitant drug medication: The following drugs cause drug interaction with S-1.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2009-04; Primary Completion 2010-10 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Disease free survival | 3 years

SECONDARY OUTCOMES:
Overall Survival | 3 years
Number of participants with adverse events as a measure of safety and tolerability | 3 year

OTHER OUTCOMES:
Health -related quality of life | 6 months after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Hee Cho, M.D.Ph.D., Principal Investigator — CNUHH
Locations (1):
- Chonnam National University Hwasun Hospital, Hwasun-Eup, Jeollanam-do, South Korea